CLINICAL TRIAL: NCT06684080
Title: A Cluster Randomized Trial on the Effectiveness of a Care Bundle to Prevent Postpartum Hemorrhage After Cesarean Delivery (Re-Team)
Brief Title: The Effectiveness of a Care Bundle to Prevent Postpartum Hemorrhage After Cesarean Delivery
Acronym: RE-TEAM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dunjin Chen (Other)
Responsible Party: Sponsor-Investigator, Dunjin Chen, Principal Investigator, The Third Affiliated Hospital of Guangzhou Medical University
Organization: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RE-TEAM
Record Dates: First submitted 2024-10-29; First posted 2024-11-12 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Cesarean Delivery
Keywords: Postpartum Hemorrhage; cesarean delivery; Randomized trial; Detection; treatment
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Care bundle group (Experimental): 1. Risk evaluation for PPH and Reserve plan; 2.Assess blood loss using Estimated Blood Loss Form and amnion fluid collection drape; 3. Satisfy any of the following conditions: i. If the estimated blood loss reaches 500ml but is less than 1000ml, and any of the following abnormal indicators are present; ii. If the estimated blood loss reaches 1000ml, no other indicators need to be considered:
  1. Lack of uterine contractions
  2. Persistent bleeding
  3. Shock index (heart rate/systolic blood pressure) was greater than 0.9 Initiate the following protocols①, ②, ③, ④
     * Maintain uterus tone (Administration of Oxytocin and second-line medications to promote uterine contraction)
       * Intravenous infusion ③ Administered tranexamic acid
         * Multi-methods and Multi-disciplinary
  Interventions: Other: A care bundle
- Usual care group (No Intervention): The usual care group does not receive a PPH risk assessment and estimates blood loss visually and used various interventions for postpartum hemorrhage in accordance with local or national guidelines.

INTERVENTIONS:
Other: A care bundle — 1. Risk evaluation for PPH and Reserve plan;
  2. Assess blood loss using Estimated Blood Loss Form and amnion fluid collection drape;
  3. Satisfy any of the following conditions: i. If the estimated blood loss reaches 500ml but is less than 1000ml, and any of the following abnormal indicators are present; ii. If the estimated blood loss reaches 1000ml, no other indicators need to be considered: 1） Lack of uterine contractions 2） Persistent bleeding 3）Shock index (heart rate/systolic blood pressure) was greater than 0.9 Initiate the following protocols①, ②, ③, ④
     * Maintain uterus tone (Administration of Oxytocin and second-line medications to promote uterine contraction)
       * Intravenous infusion ③ Administered tranexamic acid ④ Multi-methods and Multi-disciplinary
  Arms: Care bundle group

SUMMARY:
Delays in the detection or inconsistent use of effective interventions of postpartum hemorrhage can result in complications or death. We designed a cluster-randomized trial to assess a multi-component strategy for the detection and treatment of postpartum hemorrhage after cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Hospital level

  1. Public hospitals
  2. There are more than 100 cesarean deliveries per year
* Patient level

  1. Cesarean delivery
  2. Sign informed consent

Exclusion Criteria:

* Hospital level

  1. Data verification information cannot be provided
* Pregnant woman level 1. No blood routine results within 2 weeks before surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52000 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of PPH | Day 2
  defined by a calculated estimated blood loss > 1000 mL [Calculated estimated blood loss = estimated blood volume × (preoperative hematocrit - postoperative hematocrit)/preoperative hematocrit (where estimated blood volume (mL) = weight (Kg) × 85)] or red blood cell (RBC) transfusion before day 2 postpartum .

SECONDARY OUTCOMES:
mean total calculated blood loss | Day 2
  Calculated estimated blood loss = estimated blood volume × (preoperative hematocrit - postoperative hematocrit)/preoperative hematocrit (where estimated blood volume (mL) = weight (Kg) × 85)]
Estimated blood loss | postpartum 24 hours
  Estimated intraoperative and postoperative blood loss at 24 hours
Incidence of postpartum transfusion | baseline
  infusion of RBC, plasma, platelet, or cryo et al
Incidence of additional operations performed outside cesarean section | baseline
  Additional operations include B-Lnych, uterine artery suture, partial hysterectomy, hysterectomy et al
Incidence of transfer to intensive care unit | baseline
  transfer to intensive care unit
Incidence of maternal death from any cause | Up to 42 days
  maternal death from any cause
The adherence to the treatment bundle | intraoperation and postpartum 24 hours
  defined adherence to at least four core bundle elements: risk evaluation for PPH and reserve plan, maintaining uterus tone (administration of oxytocin and second-line medications to promote uterine contraction), intravenous infusion, administered tranexamic acid

IPD SHARING:
Plan to Share IPD: No